CLINICAL TRIAL: NCT04739930
Title: Prospective, Randomized, Single Blind Clinical Trial to Investigate the Impact of Autologous Bone Marrow Concentrate in Knee Osteochondral Allograft Transplantation
Brief Title: Autologous Bone Marrow Concentrate in Knee Osteochondral Allograft Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Joint Restoration Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17121805
Record Dates: First submitted 2020-12-24; First posted 2021-02-05 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Cartilage Injury

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Single Blind Clinical Trial
Who Masked: Participant
Masking Description: The control group will receive a 0.5cm sham incision over the iliac crest, but bone marrow aspiration will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone Marrow Aspiration Group (Experimental): A bone marrow aspiration will be performed from the iliac crest. The bone marrow aspirate will be processed using a bone marrow aspirate concentrate (BMAC) harvesting system. The osteochondral allograft plug will then be soaked in the BMAC for a minimum 2 minutes prior to implantation. The remaining BMAC will be placed in the defect site prior to plug implantation.
  Interventions: Procedure: Autologous bone marrow aspirate will be harvested and concentrated to a bone marrow aspirate concentrate (BMAC) containing bone marrow derived mesenchymal stem cells and delivered to site of operation
- Control (Sham Comparator): The control group will receive a 0.5cm sham incision over the iliac crest, but bone marrow aspiration will not be performed. The osteochondral allograft plug will not be soaked in BMAC prior to implantation.
  Interventions: Procedure: Control group incision

INTERVENTIONS:
Procedure: Autologous bone marrow aspirate will be harvested and concentrated to a bone marrow aspirate concentrate (BMAC) containing bone marrow derived mesenchymal stem cells and delivered to site of operation — Autologous bone marrow aspirate will be processed and concentrated to a bone marrow aspirate concentrate (BMAC) containing bone marrow derived mesenchymal stem cells and delivered to the site of operation in the treatment group
  Arms: Bone Marrow Aspiration Group
Procedure: Control group incision — 0.5cm sham incision over the iliac crest
  Arms: Control

SUMMARY:
The goal of this study is to establish if mesenchymal stem cell augmentation improves graft incorporation and to analyze the cytokine environment of the joint after osteochondral allograft transplantation (OCA) with and without intra-articular bone marrow aspirate concentrate (BMAC) injection. Information learned from this study can be used to biochemically compare treatment response and to assess emerging therapeutic options that may positively alter the biochemical environment in patients who suffer from articular cartilage disorders.

DETAILED DESCRIPTION:
Articular cartilage injuries in the knee continue to grow in number as detection and treatment options have advanced. Treatment options, including microfracture, autologous chondrocyte (cells that make cartilage) implantation, osteochondral grafting and meniscus transplantation can hopefully deter the progression of degeneration and have promise to function as disease modifying solutions. Osteochondral allograft transplantation (OCA) has emerged as a preferred method of treating large focal chondral defects as it structurally replaces the cartilage and often involved sub-chondral bone with native hyaline cartilage and bone. The results of OCA are successful with greater than 85% survival at 5-year follow-up. Failure can occur due to a lack of boney integration or low chondrocyte viability. Therefore, anything to enhance the graft augmentation process may be useful in preventing failure. The purpose of this prospective, randomized study is to determine the effect of bone marrow aspirate concentrate (BMAC) containing bone marrow derived mesenchymal stem cells on improving graft incorporation and preventing failure. The effect of BMAC on the graft and intra-articular knee environment will be evaluated using 3 techniques: computed tomography (CT) imaging, synovial fluid cytokine analysis, and serum biomarker analysis. Information learned from this study can be used to biochemically compare treatment response and to assess emerging therapeutic options that may positively alter the biochemical environment in patients undergoing osteochondral allograft transplantation.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged 18-50 with a cartilage defect indicated for treatment with osteochondral allograft

Exclusion Criteria:

* Patients with known rheumatoid arthritis, any other inflammatory arthropathy or synovial tissue disorder.
* Patients with known bipolar osteoarthritis of the knee as determined by the treating physician, greater than Kellegren-Lawrence Grade 3 on x-ray imaging
* Patient with a known infection or history of infection in the affected knee

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2023-01-12 (Actual); Study Completion 2023-01-12 (Actual)

PRIMARY OUTCOMES:
Synovial Fluid Cytokine Measurement | Up to 52 weeks
  To measure the amount of cytokines and cartilage biomarkers in the synovial fluid of patients undergoing osteochondral allograft transplantation with and without BMAC augmentation at different time points

OTHER OUTCOMES:
Radiographic analysis | Day 1, Post-operative 2 weeks, 6 weeks, 12, weeks, 24 weeks, 52 weeks
  Changes in graft status will be analysed using radiographic analysis
Computed Tomography (CT) analysis | Post-operative 24 weeks
  Changes in graft status will be analysed using Computed Tomography (CT) analysis

CONTACTS AND LOCATIONS:
Overall Officials: Adam Yanke, MD, Principal Investigator — Faculty
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT04739930/Prot_001.pdf
  • Informed Consent Form: HIPAA Form (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT04739930/ICF_000.pdf
  • Informed Consent Form: Main Consent Form (2021-01-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT04739930/ICF_002.pdf